CLINICAL TRIAL: NCT00727155
Title: Improving Quality Of Life For Chronically Ill Patients Using Education Support And Skills; A Randomized Controlled Mental Trial
Brief Title: Adjusting to Chronic Conditions Using Education Support and Skills
Acronym: ACCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Cully, Jeffrey - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H23264
Record Dates: First submitted 2008-07-29; First posted 2008-08-01 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Treatment
  Interventions: Behavioral: Adjusting to Chronic Conditions Using Education Support and Skills
- 2 (No Intervention): Waitlist

INTERVENTIONS:
Behavioral: Adjusting to Chronic Conditions Using Education Support and Skills — This psychosocial intervention uses a combination of cognitive-behavioral therapy and disease self-management techniques.
  Arms: 1

SUMMARY:
Medically ill patients with Congestive Heart Failure (CHF) and Chronic Obstructive Pulmonary Disease (COPD) are at increased risk for developing symptoms of anxiety and depression and are among the least frequent users of mental health services and treatments. To address the needs of chronically ill patients, we created a time-limited psychosocial intervention to maximize treatment benefits and improve the efficiency and ability of mental health care practitioners to provide services within medical care settings. This study is separated into two randomized study groups. The first group of participants will receive the ACCESS intervention immediately. The second group of participants will be followed for a period of 6 months. After a period of 6 months, those who continue to have symptoms of depression and/or anxiety will be offered the ACCESS intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18+;
2. Confirmation of CHF or COPD diagnosis according to medical chart review;
3. Ongoing symptoms of functional limitations due to CHF (NYHA classification of II , III, or IV as obtained by telephone interview) or COPD (Score of 3 or greater on the Medical Research Council Dyspnoea Scale [MRC] as obtained by telephone interview);
4. Eligible patients must have clinically significant symptoms of either anxiety and/or depression as measured using patient self report questionnaires. Clinical cutoff scores for depression will be based on the Beck Depression Inventory - Second Edition (scores of 14 or more) while anxiety cutoffs will be determined using the State-Trait Anxiety Inventory - trait subscale (score of 40 or greater);
5. Eligible patients will be English-speaking, as this intervention has not yet been translated to any other language.

Exclusion Criteria:

1. History of substance abuse, bipolar disorder, psychosis or active suicidal intent (obtained from standardized structured clinical interview);
2. NYHA class I, or MRC levels 1 and 2. Class 1 CHF patients and Level 1 and 2 COPD patients (by definition) will have no significantly limiting CHF or COPD symptoms. This information will be obtained through patient self-report of CHF and COPD symptoms;
3. Mental status examination score in the cognitively impaired range on an established 6-item screen;
4. Inability to provide informed consent or severe physical limitations restricting completion of the study protocol (e.g. vision, hearing, or physical functioning);
5. Non-English speaking patients will be excluded from participation, as this intervention has not yet been translated to any other language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory, State Trait Anxiety Inventory, SF-36 Health Survey | Weeks 1 (baseline), 2, 4, 6, 8, 12, 24, and 36

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Cully, PhD MEd, Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (1):
- Houston VA Medical Center, Houston, Texas, United States

REFERENCES:
- [Derived] Cully JA, Stanley MA, Deswal A, Hanania NA, Phillips LL, Kunik ME. Cognitive-behavioral therapy for chronic cardiopulmonary conditions: preliminary outcomes from an open trial. Prim Care Companion J Clin Psychiatry. 2010;12(4):PCC.09m00896. doi: 10.4088/PCC.09m00896blu. PMID 21085552